CLINICAL TRIAL: NCT02509559
Title: Effects of Propranolol (vs. Placebo) on Information Processing During Presentation of Emotionally Arousing Pictures After Single Dose (80 mg) Administration and Relationships Between ß1- and ß2-adrenoreceptors Genotype and Both the Information Processing and the Propranolol Effects in 64 Healthy Male Subjects
Brief Title: Effects of Propranolol (vs. Placebo) on Information Processing During Presentation of Emotionally Arousing Pictures
Acronym: BBEmoMem_G
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: BBEmoMem_G
Record Dates: First submitted 2015-06-30; First posted 2015-07-28 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Emotions
Keywords: Receptors, Adrenergic; Propranolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Propanolol (Active Comparator): Memory performance for pictures, electrocortical activity, pharmacokinetics, skin-conductance, pulse waves, burdening heart frequency, pulmonary function, α-amylase in saliva, heart rate and blood pressure after administration of one Propranolol-CT 80 mg film-coated tablet.
  Interventions: Drug: propranololhydrochloride; Device: Net Station® System and compatible Geodesic Sensor Nets®; Device: VITAPORT; Device: ergoselect II 100/200; Device: SpiroScout; Device: Mobil-O-Graph® PWA; Procedure: Saliva collection
- Placebo (Placebo Comparator): Memory performance for pictures, electrocortical activity, pharmacokinetics, skin-conductance, pulse waves, burdening heart frequency, pulmonary function, α-amylase in saliva, heart rate and blood pressure after administration of one placebo capsule.
  Interventions: Drug: placebo; Device: Net Station® System and compatible Geodesic Sensor Nets®; Device: VITAPORT; Device: ergoselect II 100/200; Device: SpiroScout; Device: Mobil-O-Graph® PWA; Procedure: Saliva collection

INTERVENTIONS:
Drug: propranololhydrochloride — oral administration of one capsule Propanolol-CT 80 mg Filmtabletten (propranololhydrochloride, film-coated tablet encapsulated, 80 mg, single dose) together with 240 ml tap water and blood sampling at time points blank, 15, 30, 45 min, 1, 2, 3, 4, 6, 8, 10, 12 h of study days 1 and 3 and urine sampling for 24 h at study days 1 and 3 with subsequent measuring of propranolol and its clinically relevant metabolites
  Other Names: propanolol pharmacokinetics
  Arms: Propanolol
Drug: placebo — oral administration of one placebo capsule together with 240 ml tap water and blood sampling at time points blank, 15, 30, 45 min, 1, 2, 3, 4, 6, 8, 10, 12 h of study days 1 and 3 and urine sampling for 24 h at study days 1 and 3
  Other Names: placebo capsule
  Arms: Placebo
Device: Net Station® System and compatible Geodesic Sensor Nets® — Electrocortical activity will be assessed by continuous EEG recording using Net Station® System and compatible Geodesic Sensor Nets® (Electrical Geodesics Incorporated, Eugene, OR, USA), measured at days 1, 3 and 10 of the study. Event related potentials at encoding (late positive potential, LPP) and at retrieval (ERP memory old/new effect) will be computed off-line after acquisition of the data.
Device: VITAPORT — Measurement of the skin conductance by VITAPORT (Vitaport EDV Systeme GmbH, Erftstadt, Germany) on study days 1 and 3 at the time points before administration of the study medication, during the psychophysiological measurement and at 4 h. Furthermore, the skin conductance responses will be measured on day 10 during the psychophysiological measurement.
Device: ergoselect II 100/200 — Performance of an ergometry by ergoselect II 100/200 (ergoline GmbH, Bitz, Germany) on study days 1 and 3 at 120 min. The burden will be the same wattage over 4 min, that corresponds to that of reaching 80% of the maximal heart frequency in the prestudy examination.
Device: SpiroScout — Performance of a spirometry (SpiroScout, Ganshorn Medizin Electronic GmbH, Niederlauer, Germany) with measuring of the forced expiratory volume in 1 second (FEV1) on study days 1 and 3 before administration of the study medication and at 120 min.
Device: Mobil-O-Graph® PWA — Measurement of pulse waves by Mobil-O-Graph® PWA (I.E.M., Stollberg, Germany) on study days 1 and 3 at the time points -10 min, 20, 40, 60, 80, 120 min, 3, 5, 7, 11 h.
Procedure: Saliva collection — Saliva collection will be performed on study days 1 and 3 at time points -10 min, 80 min, 120 min with subsequent measuring of the concentration of α -amylase

SUMMARY:
The main objective of the present study is to combine two lines of research, investigating the interaction between emotional processing and memory performance (on both behavioral and electrophysiological levels) and its modulation by ß-blockade.

Concerning pharmacological manipulations with ß-blockers, there are no studies, which investigated the effects of propranolol on electrophysiological (ERPs) and behavioral measures of recognition memory along with their codependence on individual variations of adrenergic receptors' polymorphisms. Till now, also the findings about genetic influences of ADRB1 and ADRB2 on recognition memory for emotional contents are lacking.

Therefore, the current investigation has been designed to replicate the former results which revealed reduced ERP correlates of recognition memory for emotional pictures due to administration of ß-blocker propranolol. Furthermore investigators goal is to test, whether there are any differences between carriers of genetic variants of the ADRB1 and ADRB2 in memory performance and/or changes in event-related potentials and in propranolol influences on the above mentioned processes.

In conclusion, investigators hypothesize: (1) a memory advantage of emotionally arousing stimuli over emotionally neutral pictures; (2) more pronounced ERP components (EPN, LPP, old-new effect) associated with encoding and memory for emotional stimuli; (3) a reduction of electrocortical correlates of emotional recognition memory (old-new effect) caused by propranolol; (4) a potential impact of genetic variants of the ADRB1 and ADRB2 on the emotional information processing and memory formation alone, and on the propranolol modulation of those processes.

Furthermore, investigators hypothesize additional pharmacodynamic effects of propranolol such as influence on skin- conductance, pulse waves, burdening heart frequency, pulmonary function and metabolomics, which might depend on the ADRB1 and ADRB2 genotype.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 35 years
* male
* caucasian
* body mass index: > 19 kg/m² and < 27 kg/m²
* genotype:

  1. being homozygote for ADRB2 haplotype 2 (variant allele) and homozygote for ADRB1 c.1165 (CC)
  2. being homozygote for ADRB2 haplotype 2 (variant allele) and homozygote for ADRB1 c.1165 (GG) or heterozygote for ADRB1 c.1165 (CG)
  3. being homozygote for ADRB2 haplotype 4 (wild-type) and homozygote for ADRB1 c.1165 (CC)
  4. being homozygote for ADRB2 haplotype 4 (wild-type) and homozygote for ADRB1 c.1165 (GG) or heterozygote for ADRB1 c.1165 (CG)
* good health as evidenced by the results of the clinical examination, ECG, ergometry and the laboratory check-up, which are judged by the clinical investigator not to differ in a clinical relevant way from the normal state; the lower limit for systolic pressure is stated with 110 mm Hg and diastolic blood pressure with 70 mmHg as well as heart frequency should not fall below 50 bpm (WHO definition)
* written informed consent

Exclusion Criteria:

* sex: female
* hepatic and renal diseases and/or pathological findings, which might interfere with pharmacokinetics and pharmacodynamics of the study medication
* existing cardiac or hematological diseases and/or pathological findings, which might interfere with the drug's safety, tolerability and/or pharmacokinetics (e.g. bradycardia, hypotonia, av- block I°)
* volunteers liable to orthostatic dysregulation, fainting, or blackouts
* peripheral circulatory disturbances
* gastrointestinal diseases and/or pathological findings (e.g. stenoses), which might interfere with pharmacokinetics and pharmacodynamics of the study medication
* obstructive disorder of breathing (e. g. asthma bronchiale)
* known allergic reactions to the active ingredients used or to constituents of the study medication
* known allergic reactions to any drug therapy in the anamnesis or actual de-allergisation
* psoriasis
* diabetes mellitus
* addiction to hypoglycemia
* pheochromocytoma
* myasthenia gravis
* drug or alcohol dependence
* positive drug or alcohol screening
* smokers of 10 or more cigarettes per day
* positive results in HIV, HBV and HCV screenings
* volunteers who are on a diet which could affect the pharmacokinetics of the drug (e. g. vegetarian
* heavy tea or coffee drinkers (more than 1L per day)
* volunteers suspected or known not to follow instructions of the clinical investigators
* volunteers who are unable to understand the written and verbal instructions, in particular regarding the risks and inconveniences they will be exposed to as a result of their participation in the study
* less than 14 days after last acute disease
* any medication within 4 weeks prior to the intended first administration of the study medication which might influence functions of the gastrointestinal tract (e.g. laxatives, metoclopramide, loperamide, antacids, H2-receptor antagonists, proton pump inhibitors, anticholinergics)
* any other medication within two weeks prior to the first administration of the study medication, but at least 10-time the half-live of the respective drug (except oral contraceptives)
* intake of grapefruit containing food or beverages within 14 days prior to administration of the study medication
* intake of poppy seed containing food or beverages within 14 days prior to administration of the study medication

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2013-10; Primary Completion 2014-02 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
hit rate | 90 min after study medication
  number of correctly recognized learned pictures over number of all pictures
false alarm rate | 90 min after study medication
  number of unlearned pictures incorrectly categorized as old over number of all pictures
dicrimination index | 90 min after study medication
  hit rate minus false alarm rate
event-related potentials (ERPs given in µV) | 90 min after study medication
  ERPs were extracted from the continuous electroencephalography signal (EEG). ERPs analyzed during encoding were late positive potentials (LPPs) in the time-range 550-1000 ms after stimulus onset. ERPs analyzed during recognition were late positive complexes (LPCs) for stimuli associated with hit responses (learned pictures correctly recognized as known) and correct rejections (unlearned pictures correctly categorized as unknown) in time range 550-700 ms after stimulus onset. Subtraction of amplitude values for both types of LPCs results in ERP old/new effects.

SECONDARY OUTCOMES:
Forced Expiratory Volume in 1 second (FEV 1) | up to 10 min before and 2 h after study medication
Skin Conductance Response (SCR in the time-window up to 6.5 s after stimulus onset, in µmho) | up to 10 min before and 90 min and 4 h after study medication
  The skin conductance will be measured between two electrodes attached to the participant's palm. SCRs will be averaged for every participant over following conditions: unpleasant, neutral and pleasant during encoding; and unpleasant old, neutral old, pleasant old, unpleasant new, neutral new, and pleasant new during recognition.
heart rate | up to 1 min before and 20, 40, 60, 80 min, 2, 3, 5, 7 and 11 h after study medication and during ergometry (0-2 min and 2-4 min) 2 h after study medication
systolic blood pressure (mmHg) | up to 1 min before and 20, 40, 60, 80 min, 2, 3, 5, 7 and 11 h after study medication and during ergometry (0-2 min and 2-4 min) 2 h after study medication
diastolic blood pressure (mmHg) | up to 1 min before and 20, 40, 60, 80 min, 2, 3, 5, 7 and 11 h after study medication and during ergometry (0-2 min and 2-4 min) 2 h after study medication
α-amylase activity in saliva | up to 1 min before and 80 min and 2 h after study medication
  concentration in U/ml
skin conductance level (SCL, in mikroSiemens over a time range of 120 s [µmho]) | up to 10 min before and 90 min and 4 h after study medication
  The skin conductance will be measured between two electrodes attached to the participant's palm.
mean arterial pressure (MAP) | up to 10 min before and 20, 40, 60, 80, 120 min, 3, 5, 7, 11 h after study medication
  It is defined as the average arterial pressure during a single cardiac cycle.

OTHER OUTCOMES:
area under the concentration time curve (AUC) of propanolol | before and 15, 30, 45, min, 1, 2, 3, 4, 6, 8, 10 and 12 h after study medication
maximum concentration (Cmax) of the concentration time curve of propanolol | before and 15, 30, 45, min, 1, 2, 3, 4, 6, 8, 10 and 12 h after study medication
time point of maximum concentration (tmax) of the concentration time curve (AUC) of propanolol | before and 15, 30, 45, min, 1, 2, 3, 4, 6, 8, 10 and 12 h after study medication
terminal half life (t1/2) of the concentration time curve of propanolol | before and 15, 30, 45, min, 1, 2, 3, 4, 6, 8, 10 and 12 h after study medication

CONTACTS AND LOCATIONS:
Overall Officials: Werner Siegmund, Prof, Principal Investigator — Department of Clinical Pharmacology
Locations (1):
- Department of Clinical Pharmacology, Ernst-Moritz-Arndt-University Greifswald, Greifswald, Mecklenburg-Vorpommern, Germany